CLINICAL TRIAL: NCT01227239
Title: A Phase I/II Study of S-1 and Oxaliplatin Combined With Radiation for Preoperative Locally Advanced Rectal Carcinoma. (SHOGUN Trial)
Brief Title: Preoperative S-1/OHP With Radiation Therapy for Low-lying Rectal Carcinoma in Neo-adjuvant Setting
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Japan Clinical Cancer Research Organization (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Toshiaki Watanabe, Teikyo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JACCRO CC-04
Record Dates: First submitted 2010-10-18; First posted 2010-10-25 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — S 1 (combination); Oxaliplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: S-1; Drug: Oxaliplatin; Radiation: Radiation

INTERVENTIONS:
Drug: S-1 — 40mg/m2 orally twice a day (BID) for 5 days a week at 1st week, 2nd week, 4th week and 5th week.
Drug: Oxaliplatin — 40-60mg/m2/week intravenously on day 1, 8, 22 and 29.
Radiation: Radiation — Total dose is 50.4Gy (1.8Gy X 28 fractions)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of S-1 and oxaliplatin combined with radiation by Phase I/II study.

The purpose of this study is as follows,

* In phase I, to determine the dose limiting toxicities (DLTs) and the maximum tolerated dose (MTD).
* In phase II, to evaluate the antitumor effect (pCR rate) and the safety .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed locally advanced and non-metastatic rectal adenocarcinoma (clinical stage T3, anyN or T4, anyN)
2. Possible to R0 resection
3. Received no prior therapy
4. Performance status (ECOG) 0-1
5. Normal organ and marrow function.
6. Sufficient oral intake

Exclusion Criteria:

1. History of serious allergic reaction
2. Patients without serious complications such as sensory neurotoxicity or serious diarrhea (with watery stool).
3. Female with pregnancy or lactation
4. Have another malignancy in the past 5 years except early stage other cancer that cure by local treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Phase I: Determine the Recommended dose (RD) | 10 weeks
  Based on the incidence of dose-limited toxicities(DLT), the RD is determined from 4 test levels
Phase II: pathological complete response rate | 12-16 week
  Pathological complete response(pCR) rate is calculated by numbers of pCR cases (grade 3) devided the number of subjected cases.

SECONDARY OUTCOMES:
R0 resection rate | 12-16 weeks
down staging rate | 12-16 weeks
local reccurence rate | 3 years
desease free survuval | 3 years
safety | 16-20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Watanabe, M.D., Principal Investigator — Tokyo University
Locations (6):
- Japan (6):
  - Nagoya University Graduate School of Medicine, Nagoya
  - Osaka Medical College, Osaka
  - Jichi Medical University Hospital, Tochigi
  - Tokyo University, Tokyo
  - Cancer Institute Hospital, Tokyo
  - Teikyo University, Tokyo

REFERENCES:
- [Derived] Ishihara S, Matsusaka S, Kondo K, Horie H, Uehara K, Oguchi M, Murofushi K, Ueno M, Mizunuma N, Shinbo T, Kato D, Okuda J, Hashiguchi Y, Nakazawa M, Sunami E, Kawai K, Yamashita H, Okada T, Ishikawa Y, Nakajima T, Watanabe T. A phase I dose escalation study of oxaliplatin plus oral S-1 and pelvic radiation in patients with locally advanced rectal cancer (SHOGUN trial). Radiat Oncol. 2015 Jan 23;10:24. doi: 10.1186/s13014-015-0333-8. PMID 25612635